CLINICAL TRIAL: NCT04045613
Title: An Open-label Multi-cohort Phase 1b/2 Study of Derazantinib and Atezolizumab in Patients With Urothelial Cancer Expressing Activating Molecular FGFR Aberrations
Brief Title: Derazantinib and Atezolizumab in Patients With Urothelial Cancer
Acronym: FIDES-02
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZB-CS-201; 2019-000359-15 (EudraCT Number)
Record Dates: First submitted 2019-07-26; First posted 2019-08-05 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Urothelial Carcinoma
Keywords: metastatic urothelial cancer; bladder cancer; Fibroblast Growth Factor Receptor; FGFR genetic aberration; targeted therapy; derazantinib; checkpoint inhibitor; immune checkpoint blockade; atezolizumab; Tecentriq; solid tumor
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Acrocephalosyndactylia | interventions — derazantinib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Substudy 1: Derazantinib 300 mg once daily (Experimental): Patients with urothelial cancer were treated with derazantinib 300 mg once daily
  Interventions: Drug: Derazantinib 300 mg once daily monotherapy
- Substudy 2 (Dose-Level 1): Derazantinib 200 mg once daily + atezolizumab 1200 mg (Experimental): Patients with any solid tumors were treated with derazantinib 200 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as intravenous (IV) infusion
  Interventions: Drug: Derazantinib 200 mg once daily + atezolizumab 1200 mg
- Substudy 2 (Dose-Level 2): Derazantinib 300 mg once daily + atezolizumab 1200 mg (Experimental): Patients with any solid tumors were treated with derazantinib 300 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Interventions: Drug: Derazantinib 300 mg once daily+ atezolizumab 1200 mg
- Substudy 3: Derazantinib 200 mg twice daily + atezolizumab 1200 mg (Experimental): Patients with urothelial cancer were treated with derazantinib 200 mg twice daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Interventions: Drug: Derazantinib 200 mg twice daily + atezolizumab 1200 mg
- Substudy 4 (Cohort 4a):Derazantinib 300 mg once daily (Experimental): Patients with FGFR inhibitor resistant urothelial cancer were treated with derazantinib 300 mg once daily
  Interventions: Drug: Derazantinib 300 mg once daily monotherapy (QD)
- Substudy 4 (Cohort 4b):Derazantinib 300 mg once daily + atezolizumab 1200 mg (Experimental): Patients with urothelial cancer were treated with derazantinib 300 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Interventions: Drug: Derazantinib 300 mg once daily + atezolizumab 1200 mg
- Substudy 5: Derazantinib 200 mg twice daily (Experimental): Patients with urothelial cancer were treated with derazantinib 200 mg twice daily
  Interventions: Drug: Derazantinib 200 mg twice daily monotherapy

INTERVENTIONS:
Drug: Derazantinib 300 mg once daily monotherapy — Derazantinib was administered orally at a dose of 300 mg once daily
  Arms: Substudy 1: Derazantinib 300 mg once daily
Drug: Derazantinib 200 mg once daily + atezolizumab 1200 mg — Derazantinib was administered orally at a dose of 200 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
  Arms: Substudy 2 (Dose-Level 1): Derazantinib 200 mg once daily + atezolizumab 1200 mg
Drug: Derazantinib 300 mg once daily+ atezolizumab 1200 mg — Derazantinib was administered orally at a dose of 300 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
  Arms: Substudy 2 (Dose-Level 2): Derazantinib 300 mg once daily + atezolizumab 1200 mg
Drug: Derazantinib 200 mg twice daily + atezolizumab 1200 mg — Derazantinib was administered orally at a dose of 200 mg twice daily in combination with atezolizumab 1200 mg every 3 weeks
  Arms: Substudy 3: Derazantinib 200 mg twice daily + atezolizumab 1200 mg
Drug: Derazantinib 300 mg once daily monotherapy (QD) — Derazantinib was administered orally at a dose of 300 mg once daily
  Arms: Substudy 4 (Cohort 4a):Derazantinib 300 mg once daily
Drug: Derazantinib 300 mg once daily + atezolizumab 1200 mg — Derazantinib was administered orally at a dose of 300 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
  Arms: Substudy 4 (Cohort 4b):Derazantinib 300 mg once daily + atezolizumab 1200 mg
Drug: Derazantinib 200 mg twice daily monotherapy — Derazantinib was administered orally at a dose of 200 mg twice daily
  Arms: Substudy 5: Derazantinib 200 mg twice daily

SUMMARY:
The purpose of this study was to evaluate efficacy of derazantinib monotherapy or derazantinib-atezolizumab in combination in patients with advanced urothelial cancer harboring fibroblast growth factor receptor (FGFR) genetic aberrations (GA) of various clinical stages of disease progression and prior treatments.

DETAILED DESCRIPTION:
The study comprised five open-label substudies (1-5) in patients with advanced urothelial cancer harboring FGFR GA (with the exception of substudy 2 which did not require a FGFR GA) who were treated by derazantinib monotherapy or derazantinib in combination with atezolizumab. The study enrolled patients with cisplatin-ineligible status, or patients whose disease progressed after either first-line treatment or prior treatment with FGFR inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed transitional cell carcinoma of the urothelium of the upper or lower urinary tract
* Recurrent or progressing stage IV disease, or surgically unresectable, recurrent or progressing disease
* Documented central FGFR genetic aberration (FGFR1, FGFR2, or FGFR3 mutations / short variants and rearrangements / fusions) (Note; Substudy 2 started with patients requiring an FGFR GA, but this requirement was removed from the protocol later on)
* Measurable disease, as defined by the Investigator using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* Adequate organ functions as indicated by Screening visit local laboratory values

Exclusion Criteria:

* Receipt of prior cancer treatment within specific interval periods
* Concurrent evidence of any clinically significant corneal or retinal disorder
* History of clinically significant cardiac disorders
* Known CNS metastases
* Concurrent uncontrolled or active infection with human immunodeficiency virus
* Active hepatitis B or chronic hepatitis B without current antiviral therapy
* Active hepatitis C
* Active tuberculosis
* Severe bacterial, fungal, viral and/or parasitic infections on therapeutic oral or IV medication at the time of first dose of study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Häckl, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (66):
- United States (7):
  - CTCA Clinical Research Inc., Atlanta, Newnan, Georgia
  - Englander Institute Weill Cornell Medicine, New York, New York
  - New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - University of Texas Southwestern Medical Center (UTSWMC), Dallas, Texas
  - MD Anderson, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - Medical Oncology Associates PS (dba Summit Cancer Centers), Spokane, Washington
- Australia (5):
  - Coastal Cancer Care, Birtinya
  - Canberra Hospital and Health Services, Canberra
  - John Flynn Private Hospital, Tugun
  - Ballarat Oncology & Haematology Services, Wendouree
  - Westmead Hospital, Westmead
- Medizinische Universitaet Wien - Allgemeines Krankenhaus der Stadt Wien (AKH) - Universitaetsklinik fuer Urologie, Vienna, Austria
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Juravinski Cancer Center, Hamilton
- Czechia (2):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni Nemocnice Olomouc, Olomouc
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre François Baclesse, Caen
  - CHU Timone / CEPCM, Marseille
  - Medical Oncology - Pitié-Salpêtrière Hopital, Paris
  - IUCT-Oncopole de Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Campus Charite Mitte, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - University Clinic Erlangen, Erlangen
  - Universitaetsklinikum Magdeburg A.oe.R, Magdeburg
  - Studienpraxis Urologie, Nürtingen
- Hungary (2):
  - National Institute of Oncology, Budapest
  - Bacs- Kiskun Megyei Korhaz, Kecskemét
- Italy (6):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IRCCS - Istituto Europeo di Oncologia IEO, Milan
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
  - ASST Valtellina e Alto Lario - UOC Oncologia Medica Ospedale di Sondrio, Sondrio
- Poland (4):
  - Wojewodzki Szpital Specjalistyczny im. Stefana Kardynala Wyszynskiego, Lublin
  - Med-Polonia Sp. z o. o., Poznan
  - Szpital Grochowski im. dr med. Rafała Masztaka Sp. z o.o., 04-073, Warszawa, Poland, Warsaw
  - Mazowiecki Szpital Onkologiczny, Wieliszew
- South Korea (11):
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Seoul St. Marys Hospital Catholic University of Korea, Seoul
- Spain (8):
  - Vall d Hebron Hospital, Barcelona
  - Hospital del Mar, Barcelona
  - IOB - Hospital Quiron Salud, Barcelona
  - ICO Hospitalet, Barcelona
  - Hospital Universitario HM Sanchinarro CIOCC, Madrid
  - Marques de Valdecilla University Hospital, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
- Switzerland (3):
  - Kantonsspital Graubünden, Chur
  - Lausanne University Hospital, Lausanne
  - UniversitaetsSpital Zuerich, Zurich
- United Kingdom (4):
  - Barts and The London School of Medicine and Dentistry - Barts Cancer Institute (BCI), London
  - The Sarah Cannon Research Institute, London
  - University College London Hospitals, London
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Necchi A, Ramlau R, Falcon Gonzalez A, Chaudhry A, Todenhofer T, Tahbaz R, Fontana E, Giannatempo P, Deville JL, Pouessel D, Yoon S, Powles T, Bernat M, Hackl M, Marszewska M, McKernan P, Saulay M, Scaleia F, Engelhardt M, Loriot Y, Siefker-Radtke A, De Santis M. Derazantinib alone and with atezolizumab in metastatic urothelial carcinoma with activating FGFR aberrations. JNCI Cancer Spectr. 2024 Apr 30;8(3):pkae030. doi: 10.1093/jncics/pkae030. PMID 38627238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August, 2019 to September, 2022, 321 patients underwent molecular screening, 131 underwent clinical screening, and 95 entered the study and were assigned treatment
Groups:
- Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg: Patients with solid tumors were treated with derazantinib 200 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as intravenous (IV) infusion
  Derazantinib 200 mg once daily + atezolizumab 1200 mg: Derazantinib was administered orally at a dose of 200 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
- Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg: Patients with solid tumors were treated with derazantinib 300 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Derazantinib 300 mg once daily + atezolizumab 1200 mg: Derazantinib was administered orally at a dose of 300 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
- Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily: Patients with urothelial cancer were treated with derazantinib 300 mg once daily
  Derazantinib 300 mg once daily monotherapy: Derazantinib was administered orally at a dose of 300 mg once daily
- Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg: Patients with urothelial cancer were treated with derazantinib 300 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Derazantinib 300 mg once daily + atezolizumab 1200 mg: Derazantinib was administered orally at a dose o f 300 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
Period: Overall Study
Arm/Group | Substudy 1: Derazantinib 300 mg Once Daily | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 5: Derazantinib 200 mg Twice Daily
Started | 32 | 14 | 12 | 2 | 8 | 10 | 17
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 32 | 14 | 12 | 2 | 8 | 10 | 17
Not completed — Adverse Event | 2 | 2 | 1 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 5 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 3 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other reasons | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease: Clinical progression | 1 | 0 | 3 | 1 | 1 | 3 | 3
Not completed — Progressive disease: Radiological progression | 24 | 6 | 8 | 0 | 6 | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily+ Atezolizumab 1200 mg: Patients with solid tumors were treated with derazantinib 200 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Derazantinib 200 mg once daily+ atezolizumab 1200 mg: Derazantinib was administered orally at a dose of 200 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
- Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily+ Atezolizumab 1200 mg: Patients with solid tumors were treated with derazantinib 300 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Derazantinib 300 mg once daily+ atezolizumab 1200 mg: Derazantinib was administered orally at a dose of 300 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
- Total: Total of all reporting groups
Arm/Group | Substudy 1: Derazantinib 300 mg Once Daily | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily+ Atezolizumab 1200 mg | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily+ Atezolizumab 1200 mg | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 5: Derazantinib 200 mg Twice Daily | Total
Number analyzed (Participants) | 32 | 14 | 12 | 2 | 8 | 10 | 17 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (10.17) | 65.6 (9.84) | 53.3 (12.58) | 67.5 (12.02) | 66.6 (11.94) | 62.7 (16.10) | 64.2 (7.61) | 64.6 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 8 | 1 | 4 | 6 | 4 | 38
  Male | 21 | 10 | 4 | 1 | 4 | 4 | 13 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 2 | 0 | 2 | 1 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  White | 18 | 12 | 5 | 2 | 2 | 7 | 12 | 58
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 9 | 1 | 5 | 0 | 3 | 2 | 4 | 24
Site of primary tumor at diagnosis [Count of Participants; unit: Participants]
  Bladder | 19 | 2 | 1 | 2 | 7 | 7 | 11 | 49
  Renal pelvis | 9 | 0 | 0 | 0 | 0 | 2 | 4 | 15
  Ureter | 3 | 0 | 1 | 0 | 1 | 1 | 2 | 8
  Missing | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other site of primary tumor | 0 | 12 | 10 | 0 | 0 | 0 | 0 | 22
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — The ECOG PS scale indicates increasing levels of disability, with 0 indicating fully active; 1, restricted in strenuous activity; 2, restricted in work activity but ambulatory and capable of self-care
  Participants
    Scale 0 | 14 | 4 | 2 | 1 | 0 | 2 | 8 | 31
    Scale 1 | 15 | 8 | 9 | 1 | 6 | 7 | 9 | 55
    Scale 2 | 3 | 2 | 1 | 0 | 2 | 1 | 0 | 9
Number of previous anti-cancer treatments [Count of Participants; unit: Participants]
  One treatment | 5 | 4 | 3 | 0 | 0 | 1 | 7 | 20
  Two treatments | 9 | 4 | 4 | 0 | 0 | 0 | 6 | 23
  Three or more treatments | 18 | 6 | 5 | 1 | 8 | 9 | 4 | 51
  No treatment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Prior immune checkpoint inhibitor treatment [Count of Participants; unit: Participants] | 26 | 1 | 4 | 0 | 8 | 10 | 12 | 61
Reason previous therapy ended [Count of Participants; unit: Participants]
  Treatment completed | 4 | 2 | 0 | 0 | 1 | 1 | 2 | 10
  Progressive disease | 23 | 10 | 12 | 0 | 6 | 8 | 12 | 71
  Toxicity | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3
  Other | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 5
  Unknown | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 5
  No previous therapy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Based on RECIST 1.1 (Substudies 1,3,4 and 5)
Description: ORR was defined as the proportion of patients who achieved a confirmed clinical response (CR) or partial response (PR) by blinded investigator central review (BICR) using the internationally recognized criteria for the radiological assessment in tumor response of solid tumors (RECIST) Version 1.1
Time Frame: From first dose up to 2 years
Population: Efficacy analyses were performed using the modified Intent-to-Treat (mITT) population: all patients who received at least one dose of derazantinib or atezolizumab, and had at least one post-baseline imaging assessment in accordance with RECIST 1.1, or documented clinical progression
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy 1: Derazantinib 300 mg Once Daily | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 5: Derazantinib 200 mg Twice Daily
Number analyzed (Participants) | 32 | 2 | 7 | 10 | 17
Percentage of participants | 9.4 [2.0 to 25.0] | 0.0 [0.0 to 84.2] | 14.3 [0.4 to 57.9] | 0.0 [0.0 to 30.8] | 5.9 [0.1 to 28.7]

2. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Derazantinib-atezolizumab in Combination Based on DLT Criteria, Safety and Efficacy Data (Substudy 2)
Description: The RP2D was determined by a joint decision taken by the Independent Data Monitoring Committee (IDMC), Investigators, and the Sponsor in reviewing the aggregate of DLT and AE data, and considering efficacy data
Time Frame: From first dose up to 2 years
Population: The safety/intent-to-treat (ITT) population consisted of all patients who received at least one dose of derazantinib or atezolizumab
Measure: Number; unit: mg
Groups:
- Substudy 2 Combined (Dose-Level 1 and 2): Derazantinib 200 or 300 Once Daily+ Atezolizumab 1200 mg: Patients with solid tumors were treated with derazantinib 200 mg or 300 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
Arm/Group | Substudy 2 Combined (Dose-Level 1 and 2): Derazantinib 200 or 300 Once Daily+ Atezolizumab 1200 mg
Number analyzed (Participants) | 26
mg | 300

3. Primary Outcome: Number of Patients With Dose-limiting Toxicities (DLTs) in Substudy 2
Description: In Substudy 2, the primary endpoint was the number of patients with DLTs. A DLT was defined as a clinically-significant adverse event (AE) or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications. Any DLT had to be a toxicity considered at least possibly related to derazantinib or the combination of derazantinib and atezolizumab
Time Frame: From first dose up to 2 years
Population: The maximum tolerated dose (MTD)-determining population included all patients enrolled in the MTD Part of each dose level who met the following minimum criteria during the DLT period:
  * received at least one dose of derazantinib and atezolizumab and has experienced a DLT;
  * received ≥ 90% of the derazantinib and atezolizumab dose, respectively, in Cycle 1 and did not experience a DLT, have been observed for ≥ 21 days following the first dose, and have been evaluated for safety
Measure: Number; unit: participants
Groups:
- Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg: Patients with solid tumors were treated with derazantinib 200 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Derazantinib 200 mg once daily + atezolizumab 1200 mg: Derazantinib was administered orally at a dose of 200 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
Arm/Group | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 5
participants | 0 | 0

4. Secondary Outcome: Disease Control Rate (DCR) Per RECIST 1.1 in All Substudies
Description: DCR was defined as the proportion of patients who achieved a confirmed clinical response (CR), partial response (PR) or stable disease (SD) by BICR using the internationally recognized criteria in accordance with RECIST Version 1.1
Time Frame: From first dose up to 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg: Patients with solid tumors were treated with derazantinib 200 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Derazantinib 200 mg once daily+ atezolizumab 1200 mg: Derazantinib was administered orally at a dose of 200 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
Arm/Group | Substudy 1: Derazantinib 300 mg Once Daily | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 5: Derazantinib 200 mg Twice Daily
Number analyzed (Participants) | 32 | 11 | 12 | 2 | 7 | 10 | 17
Percentage of participants | 18.8 [7.2 to 36.4] | 18.2 [2.3 to 51.8] | 50.0 [21.1 to 78.9] | 50.0 [1.3 to 98.7] | 28.6 [3.7 to 71.0] | 20.0 [2.5 to 55.6] | 52.9 [27.8 to 77.0]

5. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1
Description: DOR was calculated from the first date of documented tumor response (confirmed CR or PR) to the date of disease progression as assessed by BICR or death per RECIST 1.1
Time Frame: From first dose up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Substudy 1: Derazantinib 300 mg Once Daily | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily+ Atezolizumab 1200 mg | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily+ Atezolizumab 1200 mg | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 5: Derazantinib 200 mg Twice Daily
Number analyzed (Participants) | 32 | 11 | 12 | 2 | 7 | 10 | 17
months | 6.9 [NA to NA] — Value(s) could not be evaluable due insufficient number of participants with events | NA [NA to NA] — Value(s) could not be evaluable due insufficient number of participants with events | 7.4 [6.9 to 7.9] | NA [NA to NA] — Value(s) could not be evaluable due insufficient number of participants with events | 3.3 [NA to NA] — Value(s) could not be evaluable due insufficient number of participants with events | NA [NA to NA] — Value(s) could not be evaluable due insufficient number of participants with events | NA [NA to NA] — Value(s) could not be evaluable due insufficient number of participants with events

6. Secondary Outcome: ORR Based on RECIST 1.1 (Substudy 2)
Description: as for outcome 1
Time Frame: From first dose up to 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg: Patients with solid tumors were treated with derazantinib 300 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Derazantinib 300 mg once daily+ atezolizumab 1200 mg: Derazantinib was administered orally at a dose of 300 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
Arm/Group | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg
Number analyzed (Participants) | 11 | 12
Percentage of participants | 0.0 [0.0 to 28.5] | 16.7 [2.1 to 48.4]

7. Secondary Outcome: Progression-free Survival (PFS) by RECIST in All Substudies
Description: PFS was calculated as the time from cohort assignment until disease progression as assessed by BICR, or death from any cause, whichever came first
Time Frame: From first dose up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Substudy 1: Derazantinib 300 mg Once Daily | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily+ Atezolizumab 1200 mg | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 5: Derazantinib 200 mg Twice Daily
Number analyzed (Participants) | 32 | 11 | 12 | 2 | 7 | 10 | 17
months | 2.0 [1.9 to 2.1] | 2.0 [1.5 to 2.1] | 4.2 [0.7 to 10.8] | 2.5 [0.6 to 4.4] | 2.0 [0.6 to 4.7] | 1.9 [0.2 to 4.1] | 2.1 [2.1 to 7.0]

8. Secondary Outcome: Overall Survival (OS) in All Substudies
Description: OS was calculated from the date of cohort assignment until death from any cause
Time Frame: From first dose up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Substudy 1: Derazantinib 300 mg Once Daily | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily+ Atezolizumab 1200 mg | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 5: Derazantinib 200 mg Twice Daily
Number analyzed (Participants) | 32 | 11 | 12 | 2 | 7 | 10 | 17
months | 4.7 [3.4 to 7.3] | 8.7 [3.0 to NA] — Value(s) could not be evaluable due insufficient number of participants with events | 12.6 [2.5 to NA] — Value(s) could not be evaluable due insufficient number of participants with events | 4.2 [2.3 to 6.2] | NA [2.3 to NA] — Value(s) could not be evaluable due insufficient number of participants with events | 6.2 [1.1 to 11.8] | 7.5 [5.6 to 9.0]

9. Secondary Outcome: Number of Patients With at Least Grade 3 Adverse Events (AEs)
Description: Common Terminology Criteria for Adverse Events (CTCAE) displayed by increasing severity grades 3 to 5 (CTCAE grade 3/4/5 )
Time Frame: From first dose and until 90 days following the last dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily+ Atezolizumab 1200 mg: Patients with solid tumors were treated with derazantinib 200 mg once daily in combination with atezolizumab 1200 mg given every 3 weeks as IV infusion
  Derazantinib 200 mg once daily + atezolizumab 1200 mg: Derazantinib was administered orally at a dose of 200 mg once daily in combination with atezolizumab 1200 mg every 3 weeks
Arm/Group | Substudy 1: Derazantinib 300 mg Once Daily | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily+ Atezolizumab 1200 mg | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 5: Derazantinib 200 mg Twice Daily
Number analyzed (Participants) | 32 | 14 | 12 | 2 | 8 | 10 | 17
Participants
  Number of patients with only unrelated CTCAE Grade ≥3 | 11 | 5 | 7 | 0 | 2 | 5 | 3
  Number of patients with related CTCAE Grade ≥3 | 11 | 3 | 3 | 2 | 2 | 4 | 9
  Number of patients without CTCAE Grade ≥3 | 10 | 6 | 2 | 0 | 4 | 1 | 5

ADVERSE EVENTS:
Time Frame: AEs were assessed from first dose and until 90 days following the last dose
Arm/Group | Substudy 1: Derazantinib 300 mg Once Daily | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg | Substudy 5: Derazantinib 200 mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 8/32 | 3/14 | 3/12 | 1/2 | 0/8 | 4/10 | 1/17
Serious Adverse Events (participants affected / at risk) | 17/32 | 4/14 | 6/12 | 1/2 | 3/8 | 6/10 | 8/17
Other Adverse Events (participants affected / at risk) | 30/32 | 14/14 | 12/12 | 2/2 | 8/8 | 10/10 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Substudy 1: Derazantinib 300 mg Once Daily (N=32) | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg (N=14) | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg (N=12) | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg (N=2) | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily (N=8) | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg (N=10) | Substudy 5: Derazantinib 200 mg Twice Daily (N=17)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 7 | 2 | 3 | 1 | 0 | 4 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Substudy 1: Derazantinib 300 mg Once Daily (N=32) | Substudy 2 (Dose-Level 1): Derazantinib 200 mg Once Daily + Atezolizumab 1200 mg (N=14) | Substudy 2 (Dose-Level 2): Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg (N=12) | Substudy 3: Derazantinib 200 mg Twice Daily + Atezolizumab 1200 mg (N=2) | Substudy 4 (Cohort 4a):Derazantinib 300 mg Once Daily (N=8) | Substudy 4 (Cohort 4b):Derazantinib 300 mg Once Daily + Atezolizumab 1200 mg (N=10) | Substudy 5: Derazantinib 200 mg Twice Daily (N=17)
Alanine aminotransferase increased (Investigations) | 10 | 2 | 5 | 0 | 2 | 2 | 5
Amylase increased (Investigations) | 4 | 1 | 2 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 12 | 2 | 3 | 0 | 2 | 2 | 4
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 2 | 1 | 1 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 6 | 0 | 0 | 0 | 1 | 2 | 3
Blood lactate dehydrogenase increased (Investigations) | 4 | 1 | 2 | 0 | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 4 | 0 | 4 | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 4 | 1 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 1 | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 4 | 2 | 1 | 1 | 1 | 2 | 1
Platelet count decreased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 3 | 2 | 0 | 0 | 0 | 1 | 2
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 2 | 2 | 0 | 1 | 3 | 1
Lymphopenia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 3 | 2 | 0 | 0 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Central serous chorioretinopathy (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Maculopathy (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Xerophthalmia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 1 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 1 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 10 | 1 | 1 | 1 | 3 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 3 | 1 | 2 | 4 | 5
Dry mouth (Gastrointestinal disorders) | 7 | 1 | 2 | 0 | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 6 | 4 | 1 | 1 | 3 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 6 | 4 | 3 | 1 | 0 | 3 | 4
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 0 | 0 | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 3 | 3 | 1 | 1 | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0 | 2 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0 | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0 | 3 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 3
Lymphoedema (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 8 | 2 | 5 | 0 | 3 | 3 | 5
Fatigue (General disorders) | 8 | 5 | 2 | 0 | 1 | 3 | 6
Mucosal inflammation (General disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 2 | 0 | 2 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 3 | 0 | 0 | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT04045613/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT04045613/SAP_001.pdf